CLINICAL TRIAL: NCT05036070
Title: Proof-of-concept Study for a New Intraocular Lens, MODEL C0001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PCOL-103-ARPV
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Lens (Experimental): Model C0001
  Interventions: Device: Model C0001
- Control Lens (Active Comparator): Model ZCB00
  Interventions: Device: Model ZCB00

INTERVENTIONS:
Device: Model C0001 — Investigational intraocular lens replaces the natural lens removed during cataract surgery in both eyes.
  Arms: Study Lens
Device: Model ZCB00 — Control intraocular lens replaces the natural lens removed during cataract surgery in both eyes.
  Arms: Control Lens

SUMMARY:
This study is a 12-month, prospective, 2-arm (1 test & 1 control), randomized (1 test:1 control), bilateral, subject/evaluator-masked clinical investigation of the EPV IOL versus the standard TECNIS monofocal control IOL.

The study will be conducted at a minimum of one to a maximum of five sites in France, with a total of 40 evaluable subjects for the investigational lens group and 40 evaluable subjects for the control lens group participating in the sub-study. The peripheral and functional testing will be conducted on a sub-group of subjects who achieve binocular uncorrected distance visual acuity (UCDVA) of 0.2 logMAR or better and/or are able to perform the driving simulator-sickness testing as determined by patient response to the SSQ (Appendix D) at the first 1-month visit.

The eye implanted first will be considered the primary study eye (first eye). Subjects will be randomized to either the investigational IOL Model C0001 or the control IOL Model ZCB00 in both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Age of study population between 60-75 years;
* Bilateral cataracts for which cataract extraction and posterior chamber IOL implantation have been planned for both eyes;
* Cataractous lens changes, as demonstrated by best-corrected distance visual acuity (BCDVA) of 0.50 decimal or worse (6/12 or 20/40 Snellen) either with or without a glare source present (e.g., Brightness Acuity Tester) or with significant cataract-related visual symptoms in the opinion of the investigator;
* Potential postoperative best-corrected distance visual acuity (BCDVA) of 0.66 decimal (6/9 or 20/30 Snellen) or better;
* Drives a car at least 1-2 times per month;
* Corneal astigmatism:

  * Normal corneal topography
  * Predicted postoperative residual refractive cylinder based on a toric IOL calculator, taking surgically induced astigmatism (SIA) into account and using the posterior corneal astigmatism (PCA) option, must be less than 1.00 D in both eyes.
* Clear intraocular media other than cataract in each eye;
* Availability, willingness, sufficient cognitive awareness to comply with examination procedures;
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries;
* Ability to understand, read and write in French.

Exclusion Criteria:

* Requiring an intraocular lens power needed to achieve emmetropia (spherical equivalent ± 0.50 D) outside the available range of +18.0 D to +30.0 D for the Model C0001 IOL or +16.0 D to +28.0 D for the Model ZCB00 IOL;
* Pupil abnormalities (non-reactive, fixed pupils, or abnormally-shaped pupils);
* Irregular corneal astigmatism;
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject;
* Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery;
* Subjects who may be expected to require retinal laser treatment during the study;
* Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level of worse than 0.66 decimal (6/9 or 20/30 Snellen) during the study;
* Inability to achieve keratometric corneal stability preoperatively as a result of recent contact lens usage;
* Subjects with diagnosed degenerative visual disorders (e.g., retinal disorders such as macular degeneration) that are predicted to cause visual acuity losses to a level worse than 0.66 decimal (6/9 or 20/30 Snellen) during the study;
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects;
* Use of systemic or ocular medications that may affect vision;
* Prior, current, or anticipated use during the course of the study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcomes or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery);
* Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.);
* Poorly-controlled diabetes;
* Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcomes of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.); NOTE: Controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable.
* Neurological or neurodegenerative disorders that affect locomotion and cognitive function (e.g., Muscular disorders, Parkinson's disease, Alzheimer's disease etc.);
* Use of mobility aids;
* Motion Sickness Susceptibility Questionnaire Short-form (MSSQ-Short) score of ≥ 25;
* Subject has condition(s) associated with the fluctuation of hormones that could lead to refractive changes;
* Concurrent participation in any other clinical trial or participation within 30 days prior to the preoperative visit.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
MONOCULAR, PERIPHERAL REFRACTIVE ERROR | 1 month postoperative
MONOCULAR, PHOTOPIC BCDVA AT 4 M | 1 month postoperative
Adverse Events rates | 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (2):
- France (2):
  - Centre Hospitalier National d'Ophtalmologie, Paris, Île-de-France Region
  - Rothschild Foundation Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu